CLINICAL TRIAL: NCT06683001
Title: CHaracterization Of the STate of the System of Care for Patients With Chronic Heart Failure in the Regions of the Russian Federation: Identification, Diagnostics, Treatment, Observation
Brief Title: National Heart Failure Registry
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: HOSTa CHF; ХОСТА ХСН (Other: Russian equivalent)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective-retrospective observational registry of patients diagnosed with chronic heart failure in the regions of the Russian Federation.

The study is non-interventional and does not involve any interventions in clinical practice, the choice of treatment methods (including the type of medical device used and the method of surgical intervention) and examination.

A control observation group is not intended.

DETAILED DESCRIPTION:
The study will include retrospective and prospective data of patients with an outpatient or inpatient diagnosis of CHF.

The duration of the observation period of an individual patient with CHF is limited by the study period, or the patient's death, and includes the studied retrospective and dynamic prospective parameters. Prospective data of CHF (any stage and FC) subjects are planned to be included sequentially as they appear in inpatient CHF centers and outpatient CHF offices until 12/31/2027 inclusive and further upon extension of the study.

Retrospective data will be provided by chief freelance cardiologists of 33 constituent entities of the Russian Federation (Central Federal District, Ural Federal District, Siberian Federal District, Far Eastern Federal District) (individually, according to agreement)

ELIGIBILITY:
Inclusion Criteria:

* Any stage and/or any class of CHF

Exclusion Criteria:

* Subjects whose source records cant be obtained for the analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 3% of CHF subjects in the target regions of Russia will be included in that trial by performing thier medical records analysis
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Age of subjects with different phenotypes and stages of CHF | Every 12 months, up to 3 years
Female to male sex ratio of subjects with different phenotypes and stages of CHF | Every 12 months, up to 3 years
Clinical status of subjects with different phenotypes and stages of CHF | Every 12 months, up to 3 years
Proportion of employable and working subjects with different phenotypes and stages of CHF | Every 12 months, up to 3 years
The proportion of subjects with different algorithms for diagnosing CHF and the proportion of subjects with a verified diagnosis of CHF (established according to the recommended algorithm for diagnosing CHF) | Every 12 months, up to 3 years
The proportion of subjects taking drugs of each class and all four classes of the recommended four-component therapy regimen (in the overall choice and in different phenotypes of CHF; working/non-working age; working/non-working) | Every 12 months, up to 3 years
Number and proportion of subjects with wearable devices when using an online tool for identifying subjects with CHF with indications for high-tech medical care | Every 12 months, up to 3 years
Number and proportion of subjects when using an online tool for identifying subjects with CHF with indications for high-tech medical care | Every 12 months, up to 3 years

SECONDARY OUTCOMES:
Proportions of subjects with an increase in EF ≥10% and a decrease in the functional class of CHF by 1 point | Every 12 months, up to 3 years
The proportion of subjects hospitalized for decompensated CHF in the departments of therapeutic and cardiology profiles * | Every 12 months, up to 3 years
Proportion of subjects with newly diagnosed type 2 diabetes* | Every 12 months
Proportion of subjects with deterioration of renal function* | Every 12 months, up to 3 years
Proportion of subjects with newly diagnosed malignant neoplasm* | Every 12 months, up to 3 years
Proportion of subjects who died from CV causes* | Every 12 months, up to 3 years
Proportion of subjects with different causes of death* | Every 12 months, up to 3 years
Incidence and event rates (per 100 subject-years) for hospitalizations due to HF* | Every 12 months, up to 3 years
Incidence and event rates (per 100 subject-years) for death from CV causes* | Every 12 months, up to 3 years
Incidence and event rates (per 100 subject-years) for death from any cause* | Every 12 months, up to 3 years
The proportion of subjects with preferential drug provision for cardiovascular disease, diabetes mellitus* | Every 12 months, up to 3 years
Average frequency of outpatient visits of subjects with CHF to medical institutions* | Every 12 months, up to 3 years
The proportion of subjects registered with a cardiologist or therapist with different phenotypes and stages of CHF* | Every 12 months, up to 3 years
Average frequency of telephone patronage * | Every 12 months, up to 3 years
  *- in the overall sample and in groups of subjects with HFrEF, HFmrEF, HFpEF and in different age categories (18-49 years; 50-64 years; 65-74 years; 75-85 years;>85 years); of working/non-working age; employed/non-employed

CONTACTS AND LOCATIONS:
Overall Officials: Sergey A Boytsov, Prof., Study Chair — E.I.Chazov Cardiology Center; Zoya N Blankova, MD, PhD, Study Director — E.I.Chazov Cardiology Center; Fail' T Ageev, Prof., Principal Investigator — E.I.Chazov Cardiology Center
Locations (1):
- National Medical Research Center for Cardiology, Ministry of Health of Russian Federation Organization, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided